CLINICAL TRIAL: NCT00241059
Title: A Prospective, Open-label, Multicenter, International Follow-up Study on the Safety and Efficacy of Enteric-coated Mycophenolate Sodium (EC-MPS) in Kidney Transplant Recipients
Brief Title: Extension Study of the Safety and Efficacy of Enteric-coated Mycophenolate Sodium in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2405LA01E1
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, maintenance patients, tolerability, EC-MPS

ARMS (1):
- EC-MPS arm (Experimental)
  Interventions: Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
The objective of this extension study is to allow patients being treated with enteric-coated mycophenolate sodium (core study CERL080A2405LA01) to continue on the same treatment and to assess the long-term safety of EC-MPS.

ELIGIBILITY:
Inclusion Criteria:

* All patients who completed study CERL080A2405-LA01 and who are willing to continue treatment with Enteric-Coated Mycophenolate Sodium.

Exclusion Criteria:

* Other protocol-defined inclusion / exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2002-08; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Safety parameters and graft function in maintenance renal transplant recipients.

SECONDARY OUTCOMES:
Incidence of acute rejection episodes and graft survival in maintenance renal transplant recipients.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis